CLINICAL TRIAL: NCT07179770
Title: A Phase 1b Study to Assess the Effects of Belzutifan on 89Zr-DFO-girentuximab Uptake as a Surrogate to Determine CAIX Tumor Expression in Patients With Clear Cell Renal Cell Carcinoma
Brief Title: Effects of Belzutifan on 89Zr-DFO-girentuximab PET Uptake in Patients With Renal Cell Carcinoma (RCC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-01254; 5K12CA270377-02 (NIH)
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma | interventions — belzutifan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Previously treated metastatic clear cell RCC (Experimental): Patients will undergo imaging with [89Zr]Zr-DFO-girentuximab PET before and 28 days after treatment with belzutifan.
  Interventions: Drug: Belzutifan; Drug: 89Zr-DFO-girentuximab; Device: 89Zr-DFO-girentuximab PET

INTERVENTIONS:
Drug: Belzutifan — 120 mg orally daily for 28 days
  Other Names: Welireg®
Drug: 89Zr-DFO-girentuximab — 10 mg single slow intravenous (IV) administration
  Other Names: TLX250-CDx
Device: 89Zr-DFO-girentuximab PET — 89Zr-DFO-Girentuximab PET before and after 4 weeks of treatment with standard-of-care (SOC) belzutifan.

SUMMARY:
The purpose of this study is to identify changes in Carbonic Anhydrase IX (CAIX) expression induced by hypoxia-inducible factor 2 alpha (HIF-2α) inhibition by initiating belzutifan single agent therapy and imaging CAIX expression with 89Zr-DFO-girentuximab PET before and 4 weeks after initiating treatment. This will be the first study to evaluate potential changes in CAIX expression altered by belzutifan. Information gained from this study will be leveraged to develop combinations of belzutifan with CAIX targeted agents including radioimmunotherapy in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed advanced clear cell RCC
2. Radiographic disease progression to prior immune checkpoint inhibitor (ICI) therapy for RCC

   * ICI for adjuvant therapy: Patients who experienced radiographic tumor progression during or within 6 months after last dose of adjuvant ICI
   * ICI for locally advanced or metastatic disease: radiographic disease progression during or following ICI treatment in the 1st line setting
   * Minimum two previous treatment regimens but no maximum limit
3. Measurable disease per RECIST v1.1
4. Recovery to baseline or Grade1 NCI CTCAE v5.0 from toxicities related to any prior treatments, unless adverse events are clinically nonsignificant and/or stable in the opinion of the investigator.
5. Age>18 years of age
6. Karnofsky performance score ≥60%
7. Patients must have adequate organ and marrow function as defined below:

   * absolute neutrophil count ≥1,000/mcL
   * platelets ≥100,000/mcL
   * total bilirubin ≤ institutional upper limit of normal (ULN)
   * Aspartate Aminotransferase (AST) (SGOT)/Alanine Aminotransferase (ALT) (SGPT ≤3 × institutional ULN
   * creatinine ≤ institutional ULN OR
   * glomerular filtration rate (GFR) ≥60 mL/min/1.73 m2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m2

     1. Patients with abnormal test results outside the allowable range, but are not clinically significant, may still enroll with PI's review and approval.
     2. Laboratory reference values should account for potential normal variations due to race, ethnicity, age, sex, and gender identity (e.g., due to surgical and/or hormonal changes).
8. Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
9. For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
10. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
11. Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.
12. Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy.
13. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
14. Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
15. Patients who agree to use an adequate method of contraception throughout the study period, starting with the administration of 89Zr-DFO-girentuximab,
16. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia.
2. Patients who are receiving any other investigational agents.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to girentuximab.
4. Patients with uncontrolled intercurrent illness at the discretion of the investigator.
5. Pregnant women are excluded from this study because belzutifan is an agent with the potential for teratogenic or abortifacient effects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Standardized Uptake Value (SUV) max uptake on 89Zr-DFO-girentuximab PET in ccRCC lesions between baseline and 4 weeks after initiation of belzutifan treatment | Baseline, Week 4
Standardized Uptake Value (SUV) peak uptake on 89Zr-DFO-girentuximab PET in ccRCC lesions between baseline and 4 weeks after initiation of belzutifan treatment | Baseline, Week 4
Occurrence of one or more grade 3 or higher toxicities by CTCAE v5 criteria | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Minas Economides, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
As this is a single institutional trial, individual participant data (IPD) will not be shared. This study will comply with the NIH Public Access Policy, which ensures that the public has access to the published results of NIH funded research. It requires scientists to submit final peer-reviewed journal manuscripts that arise from NIH funds to the digital archive PubMed Central upon acceptance for publication.